CLINICAL TRIAL: NCT04239001
Title: Prospective, Open, One-arm Clinical Study Evaluating the Efficacy and Safety of Pegylated Recombinant Human Granulocyte Stimulating Factor in Secondary Prevention of Albumin Paclitaxel Combined With S-1 in the First-line Treatment of Advanced Pancreatic Cancer
Brief Title: Efficacy and Safety of Pegylated Recombinant Human Granulocyte Stimulating Factor in Secondary Prevention of Albumin Paclitaxel Combined With S-1 in the First-line Treatment of Advanced Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSPC -JYL-PC-01
Record Dates: First submitted 2020-01-09; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Advanced Pancreatic Cancer
Keywords: PEG-rhG-CSF
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEG-rhG-CSF (Experimental): Jin Youli(PEG-rhG-CSF): jinyouli injection was given 24 hours after the completion of intravenous infusion of albumin paclitaxel during the treatment period, 6 mg was given to patients with body weight ≥45 kg, and 3 mg was given for body weight <45 kg. Inject once every chemotherapy cycle
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — 24 hours after the completion of intravenous infusion of albumin paclitaxel during the treatment period, patients with pancreatic cancer who met the input / discharge criteria were given secondary prophylactic administration of the tested drug PEG-rhG-CSF.

SUMMARY:
A prospective, open, one-arm clinical study to evaluate the efficacy and safety of jinyouli in the first-line treatment of advanced pancreatic cancer with albumin paclitaxel combined with S-1.Chemotherapy regimen: (1) chemotherapy: albumin paclitaxel, 120mg / m2, intravenous infusion for 30 minutes, D1. S-1, taken orally after meal, D1 - 14. (2) patients who met the input / discharge criteria were given jinyouli injections 24 hours after the end of intravenous infusion of albumin paclitaxel during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18 years, ≤70 years;
* (2) Patients with Advanced Pancreatic Cancer diagnosed by histopathology，the expected survival time is more than 3 months;
* (3) Neutropenia of ≥2 degree occurred with the albumin paclitaxel + S-1 regimen in the previous cycle.
* (4) KPS score≥70points;
* (5) The peripheral blood routine of the patients was normal: ANC ≥ 2.0x109 / L, platelet count ≥ 90 × 109 / L, HB ≥ 80g / L before enrollment, and there was no bleeding tendency;
* (6) Patients volunteered to participate in the trial and signed a written informed consent to be followed up.

Exclusion Criteria:

* (1) There are currently hard-to-control infections or systemic antibiotic treatment within 72 h of chemotherapy；
* (2) Any abnormal bone marrow hyperplasia and other abnormal hematopoietic function；
* (3) Patients who had received bone marrow or hematopoietic stem cell transplantation within the previous 3 months；
* (4) Previous patients with other malignant tumors not cured, or brain metastases；
* (5) Liver function tests total bilirubin (TBIL), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) are >2.5 times the upper limit of normal, if the above indicators are >5 times due to liver metastasis Upper limit of normal value;
* (6) Renal function test: serum creatinine (Cr) exceeded the upper limit of normal value；
* (7) Allergic to this product or other biological products derived from genetically engineered escherichia coli；
* (8) Suffering from a mental or nervous system disorder, lacking self-awareness or coordination；
* (9) Patients who are expected to have a short survival and have difficulty tolerating chemotherapy；
* (10) Pregnant and nursing female patients；
* (11) People who are using other drugs of the same category or are in clinical trials of other drugs；
* (12) The investigator judges patients who are not suitable for participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of degree 3-4 neutropenia in each cycle of chemotherapy | It lasts 4 cycles(each cycle is 21 days)
  Incidence of degree 3-4 neutropenia in each cycle of chemotherapy

SECONDARY OUTCOMES:
The incidence of febrile neutropenia in each cycle of chemotherapy | It lasts 4 cycles(each cycle is 21 days)
  Febrile neutropenia (FN) is defined as oral temperature >38.3 ° C (underarm temperature >38.1 ° C) or continuous measurement of oral temperature >38 ° C (underarm temperature >37.8 ° C) in 2 h, and ANC <0.5×10^9/L, or expected to be <0.5×10^9/L
Incidence of chemotherapy dose adjustment due to neutropenia in each cycle of chemotherapy | It lasts 4 cycles(each cycle is 21 days)
  Incidence of chemotherapy dose adjustment due to neutropenia in each cycle of chemotherapy
The proportion of patients hospitalized due to neutropenia | It lasts 4 cycles(each cycle is 21 days)
  The proportion of patients hospitalized due to neutropenia
The proportion of patients receiving antibiotics during the entire chemotherapy period. | It lasts 4 cycles(each cycle is 21 days)
  The proportion of patients receiving antibiotics during the entire chemotherapy period.

CONTACTS AND LOCATIONS:
Overall Officials: Guanghai Dai, Principal Investigator — Chinese PLA General Hospital First medical center
Locations (1):
- Chinese PLA General Hospital First medical center, Beijing, China